CLINICAL TRIAL: NCT00621829
Title: Pilot Study of Supplemental Eicosapentanoic Acid (EPA)-Enriched Omega-3 Polyunsaturated Fatty Acids (n3-PUFA) in a Subset of Moderate to Severe Asthmatics With Polymorphisms of the Arachidonate 5-lipoxygenase (ALOX5) Gene
Brief Title: Fish Oil to Prevent Asthma Exacerbations in Patients With ALOX5 Polymorphisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200715569; CHNR07702 (Other: Other)
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fatty Acids, Omega-3; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): "High" susceptibility ALOX5 gene polymorphisms. Patients will be classified as having high susceptibility ALOX5 gene polymorphisms based on the number of repeats of the SP1 promoter.
  Interventions: Dietary Supplement: EPA enriched fish oils
- 2 (Active Comparator): "Low" susceptibility ALOX5 gene polymorphisms. "Low" susceptibility ALOX5 gene polymorphisms. Patients will be classified as having high susceptibility ALOX5 gene polymorphisms based on the number of repeats of the SP1 promoter.
  Interventions: Dietary Supplement: EPA enriched fish oils

INTERVENTIONS:
Dietary Supplement: EPA enriched fish oils — Subjects will take the (EPA)-enriched omega-3 polyunsaturated fatty acids (n3-PUFA) supplements as a capsule (3-4 g of EPA/day) for 90 days, followed by an 8 week washout period, and then will take a Placebo capsule for 90 days.
  Other Names: The study agent, a single-ingredient preparation,; is a commercially prepared and marketed fish oil; concentrate produced by Ocean Nutrition Canada (ONC); Limited (http://www.ocean-nutrition.com/). This supplement; and related products are sold under the MEG-3® brand.
  Arms: 1
Dietary Supplement: EPA enriched fish oils — Subjects will take a Placebo capsule for 90 days, followed by an 8 week washout period, and then will take the (EPA)-enriched omega-3 polyunsaturated fatty acids supplements as a capsule (3-4 g of EPA/day) for 90 days.
  Other Names: omega 3 fatty acids; fish oil; Eicosapentanoic acids
  Arms: 2

SUMMARY:
This is a clinical study that is designed to study the effects of the supplemental intake of enriched omega-3 polyunsaturated fatty acids (fish oil) in patients with moderate to severe asthma. Some asthmatics produce a large amount of inflammatory leukotriene proteins-proteins that contribute to wheezing and inflammation in the airway. Inhibiting the detrimental effects of leukotrienes is a key goal of controller therapy in severe asthmatics. Some asthmatic patients appear to have specific mutations of the arachidonate 5-lipoxygenase (ALOX5) gene, one gene that regulates the production of the inflammatory leukotrienes. Omega-3 fatty acids can interfere with the arachidonic acid pathway and decrease the production of leukotrienes, and this may benefit moderate and severe asthma patients. Our hypothesis is that omega-3 fatty acid supplements, added on to a patient's asthma medication regimen, can decrease the number of minor asthma exacerbations compared to patients who do not receive the supplement. Furthermore, we believe that asthma patients with specific ALOX5 gene mutations will benefit most. We will enroll 30 asthma subjects to take part in this trial. They will undergo genotyping of the ALOX5 gene and be treated with omega3-fatty acids (fish oil) and placebo over a nine month period. We expect that this strategy will allow us to discover which moderate and severe asthma patients will benefit most from supplements of omega-3 fatty acids. Treatment of chronic diseases, such as asthma, is a key mission of the Center of Health and Nutrition Research.

DETAILED DESCRIPTION:
This study is a single-center, investigator-initiated, randomized, double-blind, placebo-controlled, cross-over trial. A total of 30 subjects will be recruited from the U.C. Davis Asthma Network (UCAN) clinics. Some of the research will be conducted at the USDA-WHNRC (Western Health Nutrition Research Center) here at U.C. Davis.

This clinical trial is designed to study the effects of supplemental intake of eicosapentanoic acid (EPA)-enriched omega-3 polyunsaturated fatty acids (n3-PUFA, fish oil) in a subset of moderate to severe asthmatics, who have a high susceptibility to increased leukotriene production due to a polymorphism in the promoter region of the arachidonate 5-lipoxygenase (ALOX5) gene.

EPA competes with AA and can decrease leukotriene production; thus our central hypothesis is that EPA-enriched n3-PUFA supplements will decrease the production of inflammatory leukotrienes and decrease the number of acute exacerbations of asthma in patients with moderate to severe asthma and that these benefits will be greater in subjects with the "high susceptibility" ALOX5 promoter variants. Our specific aims are to: 1) Determine the prevalence of the "high-susceptibility" ALOX5 pathway gene polymorphisms in a diverse cohort of moderate to severe adult asthmatics, 2) Perform a 32 week (12 wk treatment A - 8 wk washout - 12 wk treatment B), blinded, cross-over design clinical trial, during which we treat 15 "high susceptibility" and 15 "low susceptibility" ALOX5 gene polymorphism asthmatics with n-3 PUFA supplements and placebo, and 3) Determine the baseline level and treatment effect of n-3 PUFA supplements on leukotriene metabolite and inflammatory cytokine production in subjects with the 'high' and 'low' susceptibility genotypes. Patients will be recruited primarily from the UC Davis Asthma Network (UCAN).

ELIGIBILITY:
Inclusion Criteria:

* Children and adults patients >18 years or older with moderate and severe asthma (as diagnosed by lung specialist physician), based on the NIH NAEPP 1997 guidelines, who do not have an acute exacerbation at the time of enrollment and are on the same asthma medications for at least 1 month

Exclusion Criteria:

* Less than 18 years of age
* Baseline FEV1 < 35% predicted
* Known or suspected allergy to fish oil products
* Pregnant women and nursing women
* Current smokers or subjects with a 20 pack-year history of smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Asthma exacerbations | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Charles Stephensen, Ph.D., Study Director — USDA, Staff Scientist; Nicholas Kenyon, MD, Principal Investigator — University of California, Davis
Locations (1):
- Ucdmc/Vanchcs Ccrc, Mather, California, United States